CLINICAL TRIAL: NCT05864885
Title: Phase I Study of Safety and Pharmacokinetics of Once-Daily Topical Solution in Male Subjects With Androgenetic Alopecia
Brief Title: Phase I Study of Safety and Pharmacokinetics of Topical Solution in Subjects With Androgenetic Alopecia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aneira Pharma, Inc. (Industry)
Collaborators: DataPharm Australia, CMAX Clinical Research, Agilex Australia (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANR C002
Record Dates: First submitted 2023-05-08; First posted 2023-05-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Androgenetic Alopecia
MeSH Terms: conditions — Alopecia | interventions — Minoxidil; Latanoprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Primary safety and pharmacokinetic data (Experimental): To obtain primary safety and pharmacokinetic data on the ANR- 001.1 when applied topically, once daily, for 7 days to the scalp
  Interventions: Drug: Minoxidil

INTERVENTIONS:
Drug: Minoxidil — Topical formulation applied once a day.
  Other Names: Latanoprost

SUMMARY:
This study will be a single center, open-label study of a single concentration of ANR- 001.1. The solution will be applied to the scalp of 14 male subjects by study staff once daily for 7 days.

DETAILED DESCRIPTION:
At screening, subjects will sign informed consent and inclusion and exclusion will be reviewed for each subject. Screening data will include demographics, medical history, concomitant medications, physical examination, weight, O2 sat, vital signs laboratory evaluation (CMP, CBC, UA), and ECG.

At Day 1, a physical exam, weight, O2 sat, vital signs (including BP, pulse, respiratory rate and temperature) and review of concomitant medications will be performed, and admission criteria reviewed.

If criteria are met, the study staff will administer the first dose of study medication to the area of hair loss on the scalp (8 cm x 6 cm). If there is no hair loss the dose will be administered to the crown of the head (8 cm x 6 cm). The study staff will continue to administer the study medication to the same area of the scalp of the subject, once daily for Study Days 1, 2, 3, 4, 5, 6, and 7. Daily subject visits will include vital signs, review of adverse events and concomitant medications. PK draws and ECGs will take place at Study Days 1, 2, 7 and 8, following the first dose and the last doses, respectively.

ELIGIBILITY:
Inclusion Criteria:

Males between age 18 to 65 years, in general good health. Good health is defined as a subject without any active diseases. Not included in active diseases are:

* Migraines
* Non-hospitalized depression o Asthma
* Cholecystectomy
* Gilbert's syndrome

  * Clinical diagnosis of AGA with grade II to VI hair loss on Norwood Hamilton Classification System
  * Subjects of any Fitzpatrick skin type or race provided their degree of skin pigmentation does not, in the Investigator's opinion, interfere with study assessments.
  * No known allergy to ANR-001.1 or any of its components.
  * Subject is willing to avoid extensive sun exposure, phototherapy, or use of tanning salon for the duration of the study.

Exclusion Criteria:

If subjects have a BMI outside of the range of 18-35kg/m2

* Subjects using a minoxidil product (e.g., Rogaine or generic Rogaine) or a latanoprost product (e.g., Xalatan or generic Xalatan) within 30 days of the start of Day 1 of the study.
* Subjects whose vital signs, ECG, safety labs or physical exam results are clinically significant in the opinion of the investigator.
* Subjects have a skin condition that, in the Investigators opinion, could interfere with study assessment or put the subject at undue risk by study participation.
* Subjects with an active or recent (within 30 days before Day 1) disease or infection, or chronic dermatological condition (eczema, psoriasis, infection, etc.).
* Subjects with known or suspected hypersensitivity or allergic reaction to any of the active or inactive components of the test treatment.
* Current enrollment in any other investigational medication (drug) study within the 4 weeks prior to study initiation.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 14 (Estimated)
Dates: Start 2023-06-09 (Estimated); Primary Completion 2023-07-17 (Estimated); Study Completion 2023-07-17 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic data: Cmax | 7 days
  Individual and mean maximum plasma concentration (Cmax)
Pharmacokinetic data: tmax | 7 days
  Individual and mean tmax
Pharmacokinetic data: Half-life (t1/2) | 7 days
  Individual and mean half-life (t1/2)
Pharmacokinetic data: AUC | 7 days
  Individual and mean area under the concentration-time curve calculated from time zero to the last observable concentration at time t (AUC0-t)
Pharmacokinetic data: Drug clearance | 7 days
  Individual and mean apparent clearance of drug from plasma
Safety : Skin TEAEs | 7 days
  Incidence of treatment-emergent adverse events related to skin irritation at the administration site
Safety: Systemic TEAEs | 7 days
  Incident of systemic treatment-emergent adverse events
Safety: Evaluation of QTs Interval Prolongation | 7 days
  Change from baseline in the frequency of marked QTc prolongation at each visit where ECG is performed

IPD SHARING:
Plan to Share IPD: No